CLINICAL TRIAL: NCT01108211
Title: Improving Low Bone Mass With Vibration Therapy for Girls With Adolescent Idiopathic Scoliosis (AIS) - A Randomized Controlled Trial
Brief Title: Improving Low Bone Mass With Vibration Therapy in Adolescent Idiopathic Scoliosis (AIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHENG Chun-yiu Jack, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VT AIS 02
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Scoliosis; Bone Diseases, Metabolic
Keywords: Adolescent Idiopathic Scoliosis; AIS; Vibration Therapy; Low bone mass; osteopenia
MeSH Terms: conditions — Scoliosis; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): This group will receive Vibration Therapy.
  Interventions: Device: Vibration Platform
- Observation Group (No Intervention): This group does not receive Vibration Therapy

INTERVENTIONS:
Device: Vibration Platform — The patients receive treatment by standing on the Vibration Platform 20 minutes a day, five days a week. The platform will deliver a vibration of 0.3g with a vertical displacement of 0.085mm at 35 Hz.
  Arms: Treatment Group

SUMMARY:
This is a prospective randomized controlled trial investigating the effect of vibration therapy on bone mineral density (BMD) and bone quality in AIS subjects suffering from osteopenia (low bone mass).

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional spinal deformity and AIS is the commonest with a high prevalence of 2-4 % in the general population. As many as 30% of AIS subjects also suffer from osteopenia which can persist and result in serious health problems later in life including vertebral collapse, fragility fractures, decreased quality of life and even mortality. In spite of this, a safe, effective and evidence-based treatment protocol for AIS-related osteopenia is not available. It remains uncertain how effective dietary advices, physical activity, Calcium and Vitamin D supplements are in this regard. On the other hand, low-magnitude high-frequency vibration therapy was shown to be effective in increasing bone mass both in animal models and in clinical trials involving elderly subjects. AIS-related osteopenia may have a different clinical behaviour. In addition, the in-vivo effect on bone quality has never been studied. We plan to carry out a scientific clinical study on the effect of vibration therapy on skeletally mature female AIS subjects with osteopenia. They are randomly allocated to either the treatment or the control group. BMD, bone micro-architectures are assessed to delineate whether vibration therapy has any therapeutic effect on improving low bone mass in osteopenic AIS subjects.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 25 year-old female patients suffering from clinically and radiologically diagnosed AIS
* more than 18 months post-menarche and Risser's sign equal to or greater than 4, and fusion of epiphyseal plate of all phalanges and metacarpals of the left hand and wrist.
* The Cobb's angle of the major structural curve is between 10 to 50 degrees (inclusive)
* Z-score BMD of less than -1

Exclusion Criteria:

* medical or musculoskeletal conditions that contraindicate or prevent the patients from receiving vibration therapy
* subjects who are not willing to comply with the treatment protocol
* subjects suffering from any medical conditions that affect bone metabolism such as hyperparathyroidism, hyperthyroidism, osteomalacia, acute or chronic renal or liver disease
* treatment with medication that affects bone metabolism such as bisphosphonate, steroid.
* pregnancy
* history of spinal operation done for scoliosis
* smokers or drinkers

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 1 year

SECONDARY OUTCOMES:
Bone micro-architecture | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tsz-ping Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong SAR, Guangdong, China

REFERENCES:
- See also: Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong — http://www.ort.cuhk.edu.hk/